CLINICAL TRIAL: NCT01053975
Title: SPIROCOR Coronary Outcome by Respiratory Stress Examination - SCORE Study
Brief Title: SPIROCOR Coronary Outcome by Respiratory Stress Examination
Acronym: SCORE
Status: Terminated | Type: Observational
Why Stopped: Based on analyses of studies separately of the SCORE study, sponsor has decided to discontinue the Study. Data collected during the study will not be analyzed
Sponsor: Spirocor (Industry)
Responsible Party: Dr. William Weintraub, Christiana Care Health Services
Other Study IDs: CM-102-005
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Severe Coronary Artery Disease (S-CAD)
Keywords: RSR; SECG; SPECT; QCA; SCAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to validate the accuracy of the SPIROCOR System in indicating the presence of significant coronary artery disease (S-CAD), as defined in ACC/AHA Guidelines, in subjects with suspected S-CAD.

ELIGIBILITY:
Inclusion Criteria:

* Subject with suspected S-CAD
* Subject able to perform the guided breathing protocol and comply with study requirements
* Subject is able and agrees to sign the informed consent form

Exclusion Criteria:

* Resting (supine) ECG evidence of ST-segment depression ≥ 1 mm in any lead or left bundle branch block or significant arrhythmia
* Current digoxin therapy
* Subject has severe valvular heart disease
* Subject has congestive heart failure NYHA class III/IV
* Subject has known history of myocardial infarction (ST elevation or non ST elevation)
* Subject had previous coronary revascularization: CABG or PCI
* Subject has pacemaker or ICD that controls sinus
* Morbidly obese subject (BMI ≥ 40)
* Subject has any significant medical condition which, at the investigator's discretion, may interfere with the subject's optimal participation in the study; and
* Subject is currently participating in another investigational product clinical study that the investigator believes may interfere with the outcome of this study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred to cardology clinics for evaluation of severe coronary artery disease (S-CAD)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
RSR vs. S-ECG in subjects suspected with S-CAD | 3 weeks window

CONTACTS AND LOCATIONS:
Overall Officials: William Weintraub, MD, Principal Investigator — Christiana Care Health Systems; Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (29):
- United States (29):
  - Cardiovascular Associates, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, Huntsville, Alabama
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Escondido Cardiology Associates, Escondido, California
  - South Denver Heart Cardiology Associates, Littleton, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Clearwater Cardiovascular & Interventional Consultants, Clearwater, Florida
  - Clearwater Cardiovascular & Interventional Consultants, Largo, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Clearwater Cardiovascular & Interventional Consultants, Safety Harbor, Florida
  - University Of Iowa Hospital, Lipid Research Clinic, Iowa City, Iowa
  - Cardiovascular Associates, Louisville, Kentucky
  - Cardiovascular Specialists of Central Maryland, PA, Columbia, Maryland
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Catholic Medical Center, Manchester, New Hampshire
  - Cardiovascular Associates of the DE Valley - Cherry Hill, Cherry Hill, New Jersey
  - Cardiovascular Associates, DE Valley- Elmer, Elmer, New Jersey
  - Cardiac & Endovascular Associates, Ridgewood, New Jersey
  - Cardiovascular Associates, DE Valley- Sewell, Sewell, New Jersey
  - Sanford Cardiology, a division of Pinehurst Medical, Inc., Sanford, North Carolina
  - The Linder Center for Research & Education, Cincinnati, Ohio
  - North Ohio Research Ltd, Elyria, Ohio
  - Humility of Mary Health Partners dba, St. Elizabeth Health Center, Youngstown, Ohio
  - Cardiac Diagnostic Associates, PC, York, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Cardiovascular Associates of East Texas, Tyler, Texas